CLINICAL TRIAL: NCT01620086
Title: Effect of Repetitive Transcranial Magnetic Stimulation (RTMS) on Resting State Brain Activity in Schizophrenia
Brief Title: Effect of Repetitive Transcranial Magnetic Stimulation on Resting State Brain Activity in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 134662
Record Dates: First submitted 2012-06-04; First posted 2012-06-15 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Auditory hallucinations (AH); Phantom sound perception; repetitive transcranial magnetic stimulation (rTMS); Percent habituation in the P50 amplitude with 250 ms ISI
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Patients with Schizophrenia who meet entry criteria for the study and first receive active repetitive transcranial magnetic stimulation for four days over a control site located at the vertex and then are randomized to receive repetitive Transcranial Magnetic Stimulation for four days over the temporal cortex at both 1 Hz and 10 Hz.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation 1 Hz; Device: Active Repetitive Transcranial Magnetic Stimulation 10 Hz; Device: Active control site Repetitive Transcranial Magnetic Stimulation at 1Hz; Device: Active control site Repetitive Transcranial Magnetic Stimulation at 10 Hz
- Controls (Experimental): These subjects are normal controls without schizophrenia who receive sham, repetitive transcranial magnetic stimulation at 1 Hz for two days and then receive active, repetitive Transcranial Magnetic stimulation for two days. All stimulation is delivered at the control site located over the vertex.
  Interventions: Device: Active control site Repetitive Transcranial Magnetic Stimulation at 1Hz; Device: Sham control site Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation 1 Hz — active rTMS delivered at 1Hz frequency over temporal cortex
  Other Names: rTMS
  Arms: Patients
Device: Active Repetitive Transcranial Magnetic Stimulation 10 Hz — active rTMS delivered at 10 Hz frequency over temporal cortex
  Other Names: rTMS
  Arms: Patients
Device: Active control site Repetitive Transcranial Magnetic Stimulation at 1Hz — active rTMS delivered at either 1 Hz frequency over the vertex
Device: Sham control site Repetitive Transcranial Magnetic Stimulation — sham rTMS delivered at 1Hz frequency over the vertex
  Arms: Controls
Device: Active control site Repetitive Transcranial Magnetic Stimulation at 10 Hz — Active 10 Hz rTMS delivered over the vertex
  Arms: Patients

SUMMARY:
This study compares the efficacy of low and high frequency repetitive transcranial magnetic stimulation (rTMS) as a means of treating subjects with schizophrenia. Magnetic pulses delivered over the scalp cause brain activity. This activity has been shown to help decrease the intensity and frequency of auditory hallucinations (AH) in schizophrenia. The investigators will compare whether low or high frequencies work best. The investigators will also examine what changes occur in the brain that are related to improvement.

DETAILED DESCRIPTION:
Background. The sub-Investigator Dr. Mennemeier has been using repetitive transcranial magnetic stimulation (rTMS) to treat phantom sound perception in subjects with tinnitus. The Principal Investigator (PI), Dr. Messias, now aims to team up with Drs. Mennemeier and James, to learn how rTMS influences phantom sound perception in schizophrenia. rTMS has already been shown to be an effective treatment for both tinnitus and schizophrenia. rTMS is a non-invasive method of regional brain stimulation that can significantly reduce phantom sound perception temporarily in 50% of subjects with tinnitus and schizophrenia. This study will go further than previous investigations by analyzing how different frequencies of rTMS influence not only auditory hallucinations (AH) in schizophrenia but also brain connectivity in schizophrenia. The investigators want to learn if rTMS decreases AH by normalizing brain connectivity. Whereas this study focuses on schizophrenic subjects with AH, the design is very similar to ongoing work on tinnitus so the findings will be comparable.

Tinnitus and AH in schizophrenia are prevalent and disabling disorders of sound perception. The investigators understanding of the precise mechanisms of these disorders is lacking. Interestingly, the symptoms of both disorders respond positively to rTMS of the temporal cortex in ways that defy contemporary understanding of the nature of these symptoms and of how rTMS should work to improve them. For example, phantom sound perception in both tinnitus and schizophrenia are linked to maladaptive, hyperactivity of auditory processing regions of temporal cortex; however, it is increasingly clear that these pathological changes alone are insufficient to explain the pronounced intrusiveness and negative emotional valance of symptoms in each disorder. Therefore, a barrier to understanding these disorders lies in understanding how changes in auditory cortex are synchronized with changes in other cortical regions that regulate perception and emotion. Additionally, at present, the decision of which rTMS frequency to apply as a treatment for phantom sound perception has no firm theoretical or empirical basis. Whereas, low frequency rTMS has traditionally been used, based upon contemporary models, to "inhibit" hyperactivity in auditory cortex; high frequency rTMS, which should induce an opposite effect on neuronal processing, not only works to improve symptoms but may be more effective for some subjects than low frequency rTMS. Therefore, contemporary models designed to explain how the frequency of rTMS influences neuronal activity immediate following stimulation are insufficient to explain how low and high frequencies of rTMS can mitigate phantom sound perception for days, weeks and months following a single course of treatment.

Hypothesis. The investigators propose that phantom sound perception in schizophrenia result from an imbalance of excitatory and inhibitory neural process in auditory networks and from synchronized, maladaptive changes in linked brain regions that regulate perception and emotion. Treating auditory cortex with repetitive, external magnetic stimulation can decrease phantom sound perception and distress by reversing the maladaptive brain reorganization that is set in motion by these underlying neural imbalances.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for schizophrenic subjects.

  * Male and female patients, 21-65 years of age, of all races and ethnicities
  * Diagnosis of auditory hallucinations (AH) associated with schizophrenia (verified at screening)
  * Must report experiencing the presence of their phantom auditory perception for at least 6 months
  * Female Subjects of childbearing age must take a pregnancy test to rule out pregnancy prior to participating in this study and during the study.
  * Willing to provide informed consent to participate in all study interventions and assessments
  * Subjects must have the capacity to sign and informed consent or a legal authorized representative (LAR) must sign in addition to the subject.
* Inclusion Criteria for control subjects.

  * Male and female patients, 21-65 years of age, of all races and ethnicities
  * Willing to provide informed consent to participate in all study interventions and assessments

Exclusion Criteria:

* Exclusion Criteria for schizophrenic subjects:

  * Subjects with significant neurological disease, acoustic neuromas or glomus tumors, or other contraindicated neuropathology.
  * Claustrophobia, or the inability to lie still in a confined space
  * Additional exclusion criteria for repetitive Transcranial Magnetic Stimulation (rTMS) include the following:

    * a personal or family history of epilepsy;
    * a personal history of head injury, aneurysm, stroke, previous cranial neurosurgery, neurological or psychiatric disorders other than schizophrenia, or migraines
    * recent use of cocaine or alcohol
    * metal implants in the head or neck
    * a pacemaker
    * pregnancy (or the possibility of pregnancy)
    * medications that lower seizure threshold (tricyclic antidepressants or bupropion) or reduce cortical excitation (anticonvulsants or benzodiazepines).
  * Persons under 21 years of age (children) are excluded because the effect of rTMS on children is unknown, in contrast to adults, who have been well studied.
  * Exclusion items specific to Functional Magnetic Resonance Imaging (fMRI):

    * magnetic metallic implants
    * electronic or magnetic implants, such as pacemakers, as these may stop working
    * nonremovable dental implants
    * permanent makeup or tattoos with metallic dyes
    * a positive pregnancy test (for females)
    * a self-reported history of loss of consciousness greater than 10 minutes
    * physical disabilities that prohibit task performance
  * Any other condition that the investigator believes might put the participant at risk
* Exclusion Criteria for control subjects:

  * Subjects with significant neurological disease, acoustic neuromas or glomus tumors, or other contraindicated neuropathology.
  * Claustrophobia, or the inability to lie still in a confined space
  * Magnetic metallic implants
  * Electronic or magnetic implants, such as pacemakers, as these may stop working
  * Nonremovable dental implants
  * Permanent makeup or tattoos with metallic dyes
  * A positive pregnancy test (for females)
  * A self-reported history of loss of consciousness greater than 10 minutes
  * Physical disabilities that prohibit task performance
  * Any other condition that the investigator believes might put the participant at risk

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erick Messias, MD, MPH, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Controls: Baseline, 1Hz Sham, 1 Hz Active Over Vertex: These subjects are normal controls without schizophrenia who receive baseline testing, then sham rTMS, and then active 1Hz rTMS. All stimulation is for two days and delivered over the control site located at the vertex.
- Patients: Baseline, Control Site, & 1Hz First: These are schizophrenic patients who meet entry criteria for the study. Patients in this arm receive baseline testing, then control site stimulation at 1Hz or 10 Hz located over the control site at the vertex, and then were randomized to receive 1 Hz over the treatment site in temporal cortex before receiving 10 Hz over the treatment site in temporal cortex. All stimulation is delivered for four days.
- Patients: Baseline, Control Site, 10Hz First: These are schizophrenic patients who meet entry criteria for the study. Patients in this arm receive baseline testing, then control site stimulation at 1Hz or 10 Hz over the control site at the vertex, and then were randomized to receive 10 Hz over the treatment site in temporal cortex before receiving 1 Hz over the treatment site in temporal cortex. All treatment is for four days.
Period: Overall Study
Arm/Group | Controls: Baseline, 1Hz Sham, 1 Hz Active Over Vertex | Patients: Baseline, Control Site, & 1Hz First | Patients: Baseline, Control Site, 10Hz First
Started | 13 | 11 | 2
Completed | 8 | 4 | 2
Not Completed | 5 | 7 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — failed study criteria | 1 | 4 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients: Patients with Schizophrenia who meet entry criteria for the study and get stimulation over temporal cortex.
- Controls: These subjects are normal controls without schizophrenia who get stimulation over the vertex.
- Total: Total of all reporting groups
Arm/Group | Patients | Controls | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.22) | 29 (9.72) | 35.2 (8.75)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Auditory Hallucinations Questionnaire (AHQ).
Description: The Auditory Hallucinations Questionnaire (AHQ) will be used to determine the patient's perceptions of change in auditory hallucinations(s). Normal controls do not fill out this measure because they do not have auditory hallucinations. Change in the average results of this test between the baseline and active treatment weeks (1 and 10 Hz) will be measured. The range of scores is 0-70, higher scores mean more symptoms.
Time Frame: change between the baseline time point and 4 days of active treatment (patients) or 2 days of sham or active treatment (controls)"
Population: Data are not collected on this outcome measure for controls. Data was missing for one patient in the active 1 Hz treatment condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Controls: 1Hz Control Site Active-Baseline; Controls: Sham Contorl Site rTMS - Baseline: These subjects are normal controls without schizophrenia.
  Baseline, no stimulation
  Active Repetitive Transcranial Magnetic Stimulation 1 Hz over vertex
  Sham Repetitive Transcranial Magnetic Stimulation at 1Hz over vertex
- Patients: Control Site-baseline; Patients: Active 1Hz Treatment Site - Baseline; Patients: Active 10 Hz Treatment Site-baseline: Patients with Schizophrenia who meet entry criteria for the study. Baseline, no stimulation
  Repetitive Transcranial Magnetic Stimulation over temporal cortex at 1 Hz
  Repetitive Transcranial Magnetic Stimulation over temporal cortex at 10 Hz
  Control site Repetitive Transcranial Magnetic Stimulation over the vertex at 1 or 10 Hz
Arm/Group | Controls: 1Hz Control Site Active-Baseline | Controls: Sham Contorl Site rTMS - Baseline | Patients: Control Site-baseline | Patients: Active 1Hz Treatment Site - Baseline | Patients: Active 10 Hz Treatment Site-baseline
Number analyzed (Participants) | 0 | 0 | 6 | 5 | 6
units on a scale |  |  | -2.67 (2.66) | -1.80 (2.86) | -2.50 (1.97)

2. Secondary Outcome: Overall Change in the Percent Habituation of the P50 Evoked Response Potential at 250 Inter Stimulus Interval (ISI) Between the Control and Active Treatments (1 and 10 Hz).
Description: Percent habituation refers to change in the amplitude of the P50 evoked response potential following a 250 ms inter stimulus interval. Change in the average results of this test between the baseline and active treatment weeks (1 and 10 Hz) will be measured.
Time Frame: as for outcome 1
Population: Three patients had missing data for the control site - baseline condition and the active 1 Hz treatment site -baseline conditions. One patient had missing data for the active 10 Hz treatment site - baseline.
Measure: Mean (Standard Deviation); unit: percent of change in wave amplitude
Arm/Group | Controls: 1Hz Control Site Active-Baseline | Controls: Sham Contorl Site rTMS - Baseline | Patients: Control Site-baseline | Patients: Active 1Hz Treatment Site - Baseline | Patients: Active 10 Hz Treatment Site-baseline
Number analyzed (Participants) | 8 | 8 | 3 | 3 | 5
percent of change in wave amplitude | -17.55 (39.17) | -6.52 (51.65) | 21 (47.63) | -23.05 (89.74) | -7.65 (68.3)

3. Secondary Outcome: Depression Level Changes as Measured by the Hamilton Depression Inventory (HAMD).
Description: HAM-D is a multiple choice questionnaire that clinicians administer to rate the severity of a subject's depression. There are 17 questions; each question has between 3-5 possible responses which increase in severity (range 0 to 52). The clinician chooses the correct response by interviewing the subject and by observing the symptoms. A score of 0-7 is considered to be normal, scores of 20 or higher indicate moderately severe depression. Change in the average results of this test between the baseline and active treatment weeks (1 and 10 Hz) will be measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls: 1Hz Control Site Active-Baseline | Controls: Sham Contorl Site rTMS - Baseline | Patients: Control Site-baseline | Patients: Active 1Hz Treatment Site - Baseline | Patients: Active 10 Hz Treatment Site-baseline
Number analyzed (Participants) | 0 | 0 | 6 | 5 | 6
units on a scale |  |  | -.083 (4.02) | -4.60 (4.88) | -3.67 (6.41)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded in a cumulative fashion for patients, and not according to the intervention received at the time of the event or according to the assigned intervention sequence.
Groups:
- Patients: These are schizophrenic patients who meet entry criteria for the study.
- Controls: These subjects are normal controls without schizophrenia.
Arm/Group | Patients | Controls
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 5/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=13) | Controls (N=13)
headache (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — headache following rTMS
sinus infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) — subject reported sinus infection
left tooth pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — left tooth and jaw pain which resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes